CLINICAL TRIAL: NCT00004373
Title: Phase II Double-Blind, Placebo-Controlled Study of the Reinforcing Effects of Alprazolam in Patients With Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11960; UTHSC-92120
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Anxiety Disorder; Panic Disorder
Keywords: anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; panic disorder; rare disease
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Alprazolam

INTERVENTIONS:
Drug: alprazolam

SUMMARY:
OBJECTIVES: I. Determine whether the benzodiazepine alprazolam reinforces self-medication behavior in anxious patients with varying histories of using other drugs.

II. Establish outpatient methods for the study of self-medication and drug reinforcement in patients vulnerable to prescription drug abuse or dependence.

III. Evaluate the influence of alcohol and other non-prescription drug use as determinants of vulnerability in these patients.

IV. Identify personality, attitudinal, or other variables that might predict different patterns of self-medication.

V. Assess the effects of cognitive-behavioral therapy on alprazolam self-medication.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This protocol involves different experiments examining self-medication with anxiolytic medications in selected patients, and cognitive-behavioral therapy for anxiety. Capsules are color coded and taken under double-blind conditions. Compliance is monitored with the Medication Event Monitoring System, which automatically registers the date and time each bottle is opened.

The physician directs therapy administration, using some combination of the following: blind choice test, antianxiety agent(s), placebo, and cognitive-behavioral therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Primary diagnosis of generalized anxiety or panic disorder Determined by Structured Clinical Interview for DSM IV
* Hamilton Anxiety Scale (HAM-A) score at least 14 AND Profile of Mood States (POMS) tension/anxiety scale score at least 20
* Concurrent diagnoses allowed: Mild to moderate agoraphobia Simple or social phobias Secondary unipolar affective disorders
* No current substance abuse, dependence, or substance abuse treatment Drug-free urine sample required
* No history of other primary Axis I diagnosis other than tobacco dependence

--Prior/Concurrent Therapy--

* No prior formalized non-drug therapy for anxiety disorder
* No concurrent prescription psychoactive medication
* No history of benzodiazepine dependence

--Patient Characteristics--

* Age: 18 to 50
* Other: Medically healthy Negative pregnancy test required No occupational requirement to work in hazardous situations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 1997-03; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: John D. Roache, Study Chair — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Roache JD, Stanley MA, Creson DR, Shah NN, Meisch RA. Alprazolam-reinforced medication use in outpatients with anxiety. Drug Alcohol Depend. 1997 May 2;45(3):143-55. doi: 10.1016/s0376-8716(97)01354-9. PMID 9179516
- [Background] Roache JD, Stanley MA: Diazepam reinforcement in anxious patients. Experimental and Clinical Psychopharmacology 4(3): 308-314, 1996.